CLINICAL TRIAL: NCT05481112
Title: Assessing Optimal XR-Buprenorphine Initiation Points in Jail
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was not initiated due to policy changes in Massachusetts (the proposed study sites).
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-00326
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Opioid Use Disorder
Keywords: XR-Buprenorphine; Sublocade; Medication for Opioid Use Disorder (MOUD)
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Sublocade

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- XR-B Induction at Admission (Experimental): Participants will initiate extended-release buprenorphine (XR-B) treatment at the time of admission. XR-B will be continued monthly from the time of induction to the day of release (up to 6 months), and up to 3 monthly injections will be offered in the community following release.
  Dosing: XR-B is available in two doses, 300mg and 100mg. Study clinicians will generally adhere to FDA-labeling on XR-B dosing, which recommends two months of 300-mg doses followed by maintenance doses of 100-mg monthly.
  Interventions: Drug: Extended-Release Buprenorphine Injection
- XR-B Induction at Pre-Release (Experimental): Participants will initiate extended-release buprenorphine (XR-B) treatment within 30 days of release. Participants will receive at least one XR-B monthly injection prior to release, and XR-B will be continued monthly from the time of induction to the day of release. Up to 3 monthly injections will be offered in the community following release.
  Dosing: XR-B is available in two doses, 300mg and 100mg. Study clinicians will generally adhere to FDA-labeling on XR-B dosing, which recommends two months of 300-mg doses followed by maintenance doses of 100-mg monthly.
  Interventions: Drug: Extended-Release Buprenorphine Injection

INTERVENTIONS:
Drug: Extended-Release Buprenorphine Injection — Extended-release buprenorphine (XR-B, Sublocade) is manufactured by Indivior. XR-B consists of a depot injectable formulation in polymeric solution to the abdomen and releases buprenorphine over 28-days (4-weeks) by diffusion as the polymer biodegrades.
  Other Names: Sublocade

SUMMARY:
The goal of this study is to compare two approaches for commencing pharmacotherapy with injectable buprenorphine for opioid use disorder (OUD) among jail inmates: (1) at the time of admission or (2) shortly before release. A sample of eligible inmates with sentences of less than 180 days will be randomly assigned to (1) initiating extended-release buprenorphine (XR-B) treatment at the time of admission (n=80), or (2) initiating XR-B treatment within 30 prior to their scheduled release date (n=80). The groups will be compared with regard to (1) how likely they were to participate in treatment, (2) levels of in-jail opioid use (via post-release interviews), (3) continuation of pharmacotherapy and other OUD treatment in the community, and (4) levels of opioid use 4 and 12 weeks following discharge (self-report and incentivized voluntary urine tests).

ELIGIBILITY:
Inclusion Criteria:

1. Incarcerated adults able to provide written informed consent in English.
2. Currently sentenced with pending release date between 3-7 months.
3. Current moderate-to-severe opioid use disorder (DSM-5)
4. Reasonable likelihood of completing 3-months or longer of community treatment (i.e., no plans to be transferred out of state or to another correctional facility)
5. Willing to accept being randomized to initiating XR-B treatment at the time of jail admission or near the time of release.

Exclusion Criteria:

1. Severe medical or psychiatric disability making participation unsafe or regular follow-up unlikely, including patients with pre-existing moderate to severe hepatic impairment are not eligible to participate
2. Pregnancy, planning conception, or breast-feeding
3. Allergy, hypersensitivity or medical contraindication to either medication
4. Chronic pain requiring opioid pain management
5. On methadone or buprenorphine (SL-B) maintenance prior to incarceration AND intending to remain on methadone or buprenorphine maintenance upon return to the community.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants who Receive XR-B within 28 Days Prior to Jail Release | Up to Month 6
  Data derived from clinic records.

SECONDARY OUTCOMES:
Proportion of Participants who Initiate Medication for Opioid Use Disorder (MOUD) during Incarceration Period | Up to Month 6
  Includes initiation of MOUD other than XR-B.
Number of Days of Opioid Use at 1 Month Post-Release | 1 Month Post-Release (Up to Month 7)
  Participants will self-report opioid use using the Timeline Followback (TLFB) method, which asks participants to estimate number of days of drug use over the previous month.
Number of Days of Opioid Use at 3 Months Post-Release | 3 Months Post-Release (Up to Month 10)
  Participants will self-report opioid use using the Timeline Followback (TLFB) method, which asks patients to estimate number of days of drug use over the previous month.
Mean Opioid Craving Visual Analogue Scale (OC-VAS) Score during Incarceration Period | Up to Month 6
  Participants indicate their level of craving for opioids by marking a 100mm visual analogue scale where 0 = no craving and 100 = maximal craving. The questionnaire is administered at baseline and then monthly over the incarceration phase.
Mean K-6 Distress Scale Score during Incarceration Period | Up to Month 6
  K-6 Distress Scale is a 6-item self-report measure of psychological distress. Participants rank each item on a 5-point Likert scale ranging from 0 (None of the time) to 4 (All of the time). The total score is the sum of responses and ranges from 0 to 24; higher scores indicate higher levels of psychological distress. The questionnaire is administered at baseline and then monthly over the incarceration phase.
Proportion of Participants who Receive a Dose of XR-B Within 28 Days after Jail Release | 1 Month Post-Release (Up to Month 7)
  Data derived from clinic records.

CONTACTS AND LOCATIONS:
Overall Officials: David Farabee, PhD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: David Farabee; david.farabee@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to data upon reasonable request. Requests should be directed to david.farabee@nyulangone.org. To gain access, data requestors will need to sign a data access agreement